CLINICAL TRIAL: NCT04203017
Title: Allogeneic Fecal Microbiota Transplantation as a Consolidation Treatment After Autologous Hematopoietic Stem Cell Transplantation in Patients With Multiple Sclerosis
Brief Title: Fecal Microbiota Transplantation After Autologous HSCT in Patients With Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: the bio-samples are corrupted for technical reasons
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Deputy Director for research, Raisa Gorbacheva Memorial Research Institute for Pediatric Oncology, Hematology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ms/fmt
Record Dates: First submitted 2019-10-30; First posted 2019-12-18 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AutoHSCT + FMT (Experimental): AutoHSCT with reduced intensity condition regimen (RIC). FMT starting D+60 up to D+120 via po capsules: 30 capsules with fecal transplant divided in two consecutive days (more accurate capsules amount is according to patients body weight)
  Interventions: Biological: allogeneic fecal microbiota

INTERVENTIONS:
Biological: allogeneic fecal microbiota — All patients receive autoHSCT with RIC (Cyclophosphamide, Antithymocyte globulin, Rituximab). After immune system reconstitution (approximately starting D+60 up to D+120), patients will receive FMT from healthy donor via po capsules.

SUMMARY:
The hypothesis of the study is that according to modern data, the pathogenesis of multiple sclerosis is inextricably linked to the patient's microbiota. Therefore, transplantation of a normal fecal microbiota (FMT) can improve the outcome of autologous hematopoietic stem cell transplantation (autoHSCT) by increasing the disease-free period and disease progression suspension for at least 5 years after transplantation, which meets the NEDA (No Evidence of Disease Activity) criteria, satisfying the current trends of clinical neurology.

DETAILED DESCRIPTION:
AutoHSCT may be a method of choice to treat patients with refractory forms of multiple sclerosis, taking into account the insufficient efficacy of first line therapy, lack of availability (government approval) and high cost of monoclonal antibodies as a second line drugs. In this setting, according to the safety-efficiency ratio the most appropriate are reduced intensity conditioning regimens in autoHSCT. In 75% of cases for refractory forms of multiple sclerosis it is possible to achieve 5 years remission with transplant mortality less than 1%. In recent years, it is quite clear that gut microbiota abnormalities may be one of mechanisms for autoimmune diseases development. Therefore, the correction of gut dysbiosis through FMT from a healthy donor can improve the effectiveness of basic therapies. Currently, FMT is a rapidly developing method of treating intestinal infections associated with multi-resistant bacteria, based on the replacement of the recipient's microbiota by the donor's microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Multiple sclerosis (Relapsing-Remitting, Secondary-Progressive, Primary-Progressive)
* AutoHSCT
* Signed informed consent
* No second tumors
* No severe concurrent illness
* 1.0-6.5 points by EDSS
* Disease duration less than 20 years
* Disease progression on 1 and/or 2 line therapy (1 point EDSS 1.0-6.0 and 0,5 point EDSS 6.0-6.5)

Exclusion Criteria:

* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
To evaluate effectiveness of autoHSCT in combination with FMT in patients with refractory multiple sclerosis | 365 days
  Multiple sclerosis progression free survival

SECONDARY OUTCOMES:
To evaluate overall survival after autoHSCT in combination with FMT in patients with refractory multiple sclerosis | 365 days
  Overall survival
To evaluate adverse effects after FMT in immunocompromised patients | 365 days
  Toxicity based NCI CTCAE ver.5.0, including analysis of severe bacterial, fungal and viral infections incidence
Quality of life status 1 | 365 days
  Multiple sclerosis-specific questionnaire - HADS (Hospital Anxiety and Depression Scale) before and after autoHSCT:
  0-7 points - normal; 8-10 - subclinically expressed anxiety/depression; 11-21 - clinically expressed anxiety/depression
Quality of life status 2 | 365 days
  Multiple sclerosis-specific questionnaire - EDSS (Expanded Disability Status Scale) before and after autoHSCT:
  0 points - Normal neurologic exam; 1.0-1.5 - No disability, minimal signs in one or two Functional Systmes (FS); 2.0-2.5 - Minimal disability in one or two FS; 3.0-3,5 - Moderate disability in one FS, fully ambulatory; 4.0-4.5 - Fully ambulatory without aid. Able to walk without aid or rest some 500 or 300 meters; 5.0-5.5 - Ambulatory without aid or rest for about 200 or 100 meters; 6.0 - Intermittent assistance required to walk about 100 meters; 6.5 - Constant bilateral assistance required to walk about 20 meters; 7.0-7.5 - Unable to walk beyond about 5 meters or more than a few steps; 8.0 - Essentially restricted to bed, but may be out of bed itself; 8.5 - Essentially restricted to bed; 9.0 - Helpless bed patient; can communicate and eat; 9.5 - Totally helpless bed patient; unable to communicate effectively or eat/swallow; 10 - Death due to MS
Evaluation of Immune system reconstitution after autoHSCT 1 | 365 days
  CD4+/CD8+ x10^9/l level before and after autoHSCT + FMT
Evaluation of Immune system reconstitution after autoHSCT 2 | 365 days
  Regulatory T-cells (CD4+CD25+CD127low, cell/mm^3) level before and after autoHSCT + FMT
Impact of autoHSCT on brain structure anatomy | 365
  MRI 3 Tesla

CONTACTS AND LOCATIONS:
Overall Officials: Boris Afanasyev, Professor, Principal Investigator — Pavlov First Saint Petersburg State Medical University
Locations (1):
- Pavlov First Saint-Petersburg State Medical University, Saint Petersburg, Russia